CLINICAL TRIAL: NCT01415349
Title: A Phase 1, Open-label, Randomized, 2-period Crossover Drug Interaction Study in Healthy Adult Subjects to Evaluate the Effect of the Proton Pump Inhibitor Omeprazole on the Pharmacokinetics of SSP-002358
Brief Title: SSP-002358 Drug Interaction Study With Omeprazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SPD557-101; 2011-001565-41 (EudraCT Number)
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Results first posted 2012-07-06 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Healthy
MeSH Terms: interventions — revexepride; Omeprazole

ARMS (2):
- SSP-002358 alone (Experimental)
  Interventions: Drug: SSP-002358
- SSP-002358 + omeprazole (Experimental): SSP-002358 + omeprazole
  Interventions: Drug: SSP-002358 + omeprazole

INTERVENTIONS:
Drug: SSP-002358 — 1 mg, oral, once
  Arms: SSP-002358 alone
Drug: SSP-002358 + omeprazole — SSP-002358 (1 mg) + omeprazole (40 mg) given orally, once
  Arms: SSP-002358 + omeprazole

SUMMARY:
This is a drug interaction study evaluating whether blood plasma concentrations of SSP-002358-base are altered when SSP-002358 is taken together with omeprazole.

ELIGIBILITY:
Inclusion criteria:

1. Age 18-55 years inclusive at the time of consent.
2. Subject is willing to comply with any applicable contraceptive requirements of the protocol and is:

   * Male, or
   * Non-pregnant, non-lactating female
   * Females must be at least 90 days post-partum or nulliparous.

Exclusion criteria:

1. Any current or recurrent disease (eg, cardiovascular, renal, liver, gastrointestinal, malignancy or other conditions) that could affect the action, absorption, or disposition of the investigational product, or could affect clinical or laboratory assessments.
2. Any known or suspected intolerance or hypersensitivity to the investigational product or omeprazole, closely related compounds, or any of the stated ingredients.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2011-08-11 (Actual); Primary Completion 2011-09-28 (Actual); Study Completion 2011-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- PRA International, Zuidlaren, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- SSP-002358 First: A single dose of 1 mg SSP-002358 in treatment period 1, a washout period, then a single dose of 1 mg SSP-002358 + a single dose of 40 mg Omeprazole in treatment period 2
- SSP-002358 + Omeprazole First: A single dose of 1 mg SSP-002358 + a single dose of 40 mg Omeprazole in treatment period 1, a washout period, then a single dose of 1 mg SSP-002358 in treatment period 2
Period: Treatment Period 1
Arm/Group | SSP-002358 First | SSP-002358 + Omeprazole First
Started | 21 | 21
Completed | 21 | 19
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Treatment Period 2
Arm/Group | SSP-002358 First | SSP-002358 + Omeprazole First
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Safety Analysis Set: Safety Analysis Set defined as all subjects who took at least 1 dose of investigational product and had at least 1 post-dose safety assessment.
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.4 (10.52)
Age, Customized [Count of Participants; unit: Participants]
  Between 18 and 55 years | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 19
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 42

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) for SSP-002358
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administrated.
Time Frame: Assessed over 48 hours post-dose
Population: Pharmacokinetic Analysis Set defined as all subjects in the Safety Analysis Set for whom the primary pharmacokinetic data were considered sufficient and interpretable. Subjects who vomited or experienced significant diarrhea between dosing and 10 hours post-dose were excluded from the pharmacokinetic descriptive statistics and statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- SSP-002358 Alone: All subjects that received only SSP-002358
- SSP-002358 + Omeprazole: All subjects that received SSP-002358 + Omeprazole
Arm/Group | SSP-002358 Alone | SSP-002358 + Omeprazole
Number analyzed (Participants) | 36 | 38
ng/ml | 3.89 (1.30) | 4.12 (1.29)
Statistical Analysis 1: Comparison: SSP-002358 Alone vs SSP-002358 + Omeprazole; Test type: Non-Inferiority or Equivalence — Point estimates and 90% confidence intervals were assessed against the currently accepted bioequivalence criteria for log-transformed data (0.80, 1.25); Mixed Models Analysis; Ratio of Geometric LS Means = 1.03, 90% CI 2-sided [0.966 to 1.09]

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity (AUC 0→∞) for SSP-002358
Description: Area under the plasma concentration versus time curve from time 0 to infinity. AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: Assessed over 48 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | SSP-002358 Alone | SSP-002358 + Omeprazole
Number analyzed (Participants) | 36 | 38
ng*h/ml | 23.3 (6.33) | 24.6 (6.31)
Statistical Analysis 1: Comparison: SSP-002358 Alone vs SSP-002358 + Omeprazole; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Ratio of Geometric LS Means = 1.04, 90% CI 2-sided [0.998 to 1.08]

ADVERSE EVENTS:
Description: Safety Analysis Set defined as all subjects who took at least 1 dose of investigational product and had at least 1 post-dose safety assessment.
Arm/Group | SSP-002358 Alone | SSP-002358 + Omeprazole
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/42
Other Adverse Events (participants affected / at risk) | 37/40 | 38/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SSP-002358 Alone (N=40) | SSP-002358 + Omeprazole (N=42)
Abdominal distention (Gastrointestinal disorders) | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Diarrhea (Gastrointestinal disorders) | 21 | 26
Flatulence (Gastrointestinal disorders) | 4 | 2
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 7 | 4
Nausea (Gastrointestinal disorders) | 6 | 13
Catheter site related reaction (General disorders) | 2 | 2
Dizziness (Nervous system disorders) | 2 | 3
Headache (Nervous system disorders) | 30 | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.